CLINICAL TRIAL: NCT03467646
Title: Long-term Follow up After Sleeve Gastrectomy Versus Roux-en-Y Gastric Bypass Versus One-Anastomosis Gastric Bypass: A Comparative Study of Weight Loss
Brief Title: Long-term Follow up After SG vs RYGB vs OAGB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Head of Bariatric Surgery Unit. Hospital general Elche, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRJC-CTO18
Record Dates: First submitted 2018-03-10; First posted 2018-03-16 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sleeve Gastrectomy (Active Comparator): Patients undergo a laparoscopic sleeve gastrectomy as bariatric procedure
  Interventions: Procedure: Sleeve Gastrectomy
- Roux-en-Y gastric bypass (Active Comparator): Patients undergo a laparoscopic Roux-en-Y gastric bypass as bariatric procedure
  Interventions: Procedure: Roux-en-Y gastric bypass
- One-Anastomosis gastric bypass (Experimental): Patients undergo a laparoscopic One-Anastomosis gastric bypass as bariatric procedure
  Interventions: Procedure: One-Anastomosis Gastric Bypass

INTERVENTIONS:
Procedure: Sleeve Gastrectomy — The patients undergo a Sleeve Gastrectomy as bariatric procedure
  Arms: Sleeve Gastrectomy
Procedure: Roux-en-Y gastric bypass — The patients undergo a Roux-en-Y gastric bypass as bariatric procedure
  Arms: Roux-en-Y gastric bypass
Procedure: One-Anastomosis Gastric Bypass — The patients undergo a One-Anastomosis Gastric Bypass as bariatric procedure
  Arms: One-Anastomosis gastric bypass

SUMMARY:
A prospective randomized clinical study of all morbidly obese patients undergoing SG, RYGB and OAGB, as primary bariatric procedures, was performed. Patients were randomly assigned into 3 groups: those patients undergoing SG, those ones undergoing RYGB and those ones undergoing OAGB. BMI, excess BMI loss (EBMIL) and remission of type 2 diabetes (T2DM), hypertension (HT) and dyslipidemia (DL) were assessed.

DETAILED DESCRIPTION:
A prospective randomized clinical study of all morbidly obese patients undergoing SG, RYGB and OAGB, as primary bariatric procedures, was performed. Patients were randomly assigned into 3 groups: those patients undergoing Sleeve Gastrectomy, those ones undergoing Roux-en-Y Gastric Bypass and those ones undergoing One-Anastomosis Gastric Bypass. Body Mass Index (BMI), excess BMI loss (EBMIL) and remission of type 2 diabetes (T2DM), hypertension (HT) and dyslipidemia (DL) were assessed.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) >40 Kg/m2
* BMI > 35 Kg/m2 with the presence of comorbidities associated to obesity
* age older than 18 years
* Patients willing to participate in the study and giving their written consent

Exclusion Criteria:

* patients undergoing other bariatric techniques than SG, RYGB and OAGB
* Patients undergoing any other surgical procedure added to the bariatric surgery
* patients with medical or surgical pathologies that at the discretion of the investigators do not allow their participation in the study
* inability to understand the nature and purpose of the study and / or to accept written participation in the study
* impossibility to comply with pre-established clinical follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Weight loss | 1 , 2 and 5 years after surgery
  The postoperative weight loss is investigated at 1, 2 and 5 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Angel Carbajo, Study Director — Centro de Tratamiento de la Obesidad

REFERENCES:
- [Derived] Ruiz-Tovar J, Carbajo MA, Jimenez JM, Castro MJ, Gonzalez G, Ortiz-de-Solorzano J, Zubiaga L. Long-term follow-up after sleeve gastrectomy versus Roux-en-Y gastric bypass versus one-anastomosis gastric bypass: a prospective randomized comparative study of weight loss and remission of comorbidities. Surg Endosc. 2019 Feb;33(2):401-410. doi: 10.1007/s00464-018-6307-9. Epub 2018 Jun 25. PMID 29943058 (Retraction: PMID 33452565 Surg Endosc. 2021 Mar;35(3):1492)